CLINICAL TRIAL: NCT03032705
Title: Clinical Evaluation of Kerr SonicFill™ 2 vs 3M ESPE Filtek™ Supreme Ultra Universal Restorative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: KaVo Kerr (Industry)
Responsible Party: Principal Investigator, Dr. Gerard Kugel, Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12311
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Results first posted 2021-11-12 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries
Keywords: Restorations; Composite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SonicFill™ 2 (Experimental): Composite: SonicFill™ 2; Bonding Agent: Optibond XRT
  Interventions: Device: SonicFill™ 2
- Filtek™ Supreme (Active Comparator): Composite: Filtek™ Supreme Ultra Universal Restorative; Bonding Agent: Scotchbond™ Universal Adhesive
  Interventions: Device: Filtek™ Supreme

INTERVENTIONS:
Device: SonicFill™ 2 — The intervention in arm 1 is SonicFill™ 2, a sonic-activated, bulk fill dental composite system for posterior restorations that requires no additional capping layer.
  Arms: SonicFill™ 2
Device: Filtek™ Supreme — The intervention in arm 2 is Filtek™ Supreme Ultra, a Universal Nanocomposite dental restorative material that is visible-light activated and designed for use in anterior and posterior restorations of any class.
  Arms: Filtek™ Supreme

SUMMARY:
The purpose of this study is to compare esthetic, functional and biological properties of two restoration materials used to fill cavities. One material is called "Filtek™ Supreme" which is a traditional tooth colored resin composite that is placed in the cavity in layers and hardened with UV light. The second material is called "SonicFill™ 2," which is a bulk fill composite that uses an ultrasonic hand piece to change the material from a solid into a liquid in order to place it into the cavity. This material can be placed in the cavity in 1 layer, and is hardened using UV light. Both materials have been FDA approved as non-significant risk devices for filling cavities.

In each subject, one tooth with a cavity will be randomly selected to receive one filling material, and a second tooth with a cavity will be randomly selected to receive the second material. The fillings will be observed over a two year period to determine clinical acceptability.

DETAILED DESCRIPTION:
This study is a randomized, split-mouth, controlled, examiner-blinded clinical evaluation of Class II restorations using a new bulk-fill composite (SonicFill™ 2) and comparing it to Filtek™ Supreme resin composite placed in the traditional incremental technique.

The primary objective of this study is to evaluate the clinical performance of a sonic-activated, bulk fill composite, SonicFill™ 2, by comparing it to Filtek™ Supreme in the following categories:

Esthetic Properties

* Surface luster
* Staining - surface
* Staining - margin
* Color match and translucency
* Esthetic anatomical form

Functional Properties

* Fracture of material and retention
* Marginal adaptation
* Approximate anatomical form - contact point
* Radio-graphic examination (when applicable)
* Patient's view

Biological Properties

* Postoperative (hyper-)sensitivity and tooth vitality
* Recurrence of caries, erosion, abfraction
* Tooth integrity (enamel cracks, tooth fractures)
* Adjacent mucosa

The hypothesis to be tested is that the sonic-activated, bulk fill composite, SonicFill™ 2, will have comparable results to the traditional incremental technique composite, Filtek™ Supreme, in overall clinical acceptability and in all compared categories

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Is willing to provide voluntary written informed consent
* Is in good medical health and able to tolerate the dental procedures
* Has at least 1 pair of qualifying molars or premolars that require Class II restorations.
* Restorations must have a buccal to lingual/palatal width equal to or greater than 1/3 the distance from buccal to lingual/palatal cusp tips
* Study teeth must be in occlusal function and must also be in contact with the neighboring tooth on at least one surface
* Study teeth must be vital (i.e., free of clinical signs and symptoms of periapical pathology)

Exclusion Criteria:

* Is currently taking part in an evaluation of other dental restorative materials
* Has chronic periodontitis or rampant caries
* Teeth exhibiting clinical signs of periapical pathology
* Teeth with a history of self-reported preoperative pulpal problems
* Women who are pregnant (self-reported). It is standard of care to post-pone routine dental procedures and radiographed until after pregnancy.
* Women who are breast feeding.
* Known allergy to resin composites or local anesthetics.
* Abnormal oral soft tissue findings (e.g., open sores, lesions)
* An employee of the sponsor or members of their immediate family.
* Condition affecting salivary flow (e.g., salivary gland disorder, Sjögren's Syndrome)
* Any restorative treatment of the teeth involved in the study in the last 12 months.
* Are unwilling or unable to have dental radiographs or photographs taken of their dentition and soft tissues
* Any other condition which is the view of the investigator may affect the ability of a patient to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kugel, DMD, MS, PhD, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unit = Teeth. 51 participants were randomized in this study, and a total of 102 teeth were studied. Therefore 51 participants and 102 units.
Units Other Than Participants: teeth
Period: Overall Study
Arm/Group | SonicFill™ 2 | Filtek™ Supreme
Started (Each participant was analyzed for both groups therefore the total number of participants is equal to participants in both groups, not the sum of both groups which is 51. Each participants contributed 2 randomly selected teeth for each study group therefore 1 participant contributing 2 study teeth in each case.) | 51; 51 teeth (Number of participants are same (repeated) for both groups unit = teeth) | 51; 51 teeth (Number of participants are same (repeated) for both groups unit = teeth)
Completion of Restorations (V2) (45 participants total for both groups) | 45; 45 teeth (Number of participants are same (repeated) for both groups unit = teeth) | 45; 45 teeth (Number of participants are same (repeated) for both groups unit = teeth)
Completed (Completion of 18 month follow up visit (Visit #5) 29 participants for SonicFill2 group 28 particiants for Filtek Supreme group) | 29; 29 teeth (Number of participants are same (repeated) for both groups unit = teeth) | 28; 28 teeth (Number of participants are same (repeated) for both groups unit = teeth)
Not Completed | 22; 22 teeth | 23; 23 teeth
Not completed — Lost to Follow-up | 16 | 17
Not completed — did not quality | 6 | 6

BASELINE CHARACTERISTICS:
Population: Each participants contributed 2 randomly selected teeth for each study group therefore 1 participant contributing 2 study teeth in each case. Therefore total number of participants is 45 and total number of units is 90.
Units Other Than Participants: teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | SonicFill™ 2 | Filtek™ Supreme | Total
Number analyzed (Participants) | 45 | 45 | 45
Number analyzed (teeth) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 43 | 86
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.13 (1.92) | 44.13 (1.92) | 44.13 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Esthetic Properties: Number of Teeth, Rated 1 (Most Desirable Outcome) to 5 (Least Desirable Outcome), in Each Esthetic Category
Description: The following properties will be evaluated using the Hickel Grading Criteria:
  1. Surface luster
  2. Staining - surface
  3. Staining - margin
  4. Color match and translucency
  5. Esthetic anatomical form
  Each criteria will be graded by blinded examiner in 5 point scale from 1 being excellent to 5 being clinically unacceptable
Time Frame: From Baseline up to 2 Years After Restoration Placement
Population: 45 Participants, each with 2 "units" (teeth) sampled. Due to participant drop out and replaced restorations, end-of-study categories have fewer than 45 units analyzed. 29 participants completed Visit 5 of the study - 28 teeth with SonicFill™ 2 (1 restoration replaced) and 27 teeth with Filtek™ Supreme (2 restorations replaced).
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | SonicFill™ 2 | Filtek™ Supreme
Number analyzed (Participants) | 45 | 45
Number analyzed (Teeth) | 45 | 45
Teeth
  Surface Luster at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Surface Luster at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Surface Luster at end of study : Number of teeth rated 1 | 25 | 25
  Surface Luster at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Surface Luster at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Surface Luster at end of study : Number of teeth rated 2 | 2 | 2
  Surface Luster at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Surface Luster at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Surface Luster at end of study : Number of teeth rated 3 | 0 | 0
  Surface Luster at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Surface Luster at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Surface Luster at end of study : Number of teeth rated 4 | 1 | 0
  Surface Luster at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Surface Luster at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Surface Luster at end of study : Number of teeth rated 5 | 0 | 0
  Surface Staining at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Surface Staining at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Surface Staining at end of study : Number of teeth rated 1 | 26 | 22
  Surface Staining at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Surface Staining at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Surface Staining at end of study : Number of teeth rated 2 | 1 | 3
  Surface Staining at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Surface Staining at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Surface Staining at end of study : Number of teeth rated 3 | 1 | 2
  Surface Staining at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Surface Staining at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Surface Staining at end of study : Number of teeth rated 4 | 0 | 0
  Surface Staining at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Surface Staining at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Surface Staining at end of study : Number of teeth rated 5 | 0 | 0
  Marginal Staining at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Marginal Staining at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Marginal Staining at end of study : Number of teeth rated 1 | 25 | 24
  Marginal Staining at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Marginal Staining at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Marginal Staining at end of study : Number of teeth rated 2 | 2 | 3
  Marginal Staining at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Marginal Staining at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Marginal Staining at end of study : Number of teeth rated 3 | 1 | 0
  Marginal Staining at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Marginal Staining at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Marginal Staining at end of study : Number of teeth rated 4 | 0 | 0
  Marginal Staining at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Marginal Staining at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Marginal Staining at end of study : Number of teeth rated 5 | 0 | 0
  Color Match and Translucency at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Color Match and Translucency at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Color Match and Translucency at end of study : Number of teeth rated 1 | 21 | 17
  Color Match and Translucency at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Color Match and Translucency at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Color Match and Translucency at end of study : Number of teeth rated 2 | 7 | 9
  Color Match and Translucency at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Color Match and Translucency at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Color Match and Translucency at end of study : Number of teeth rated 3 | 0 | 1
  Color Match and Translucency at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Color Match and Translucency at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Color Match and Translucency at end of study : Number of teeth rated 4 | 0 | 0
  Color Match and Translucency at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Color Match and Translucency at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Color Match and Translucency at end of study : Number of teeth rated 5 | 0 | 0
  Esthetic Anatomical Form at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Esthetic Anatomical Form at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Esthetic Anatomical Form at end of study : Number of teeth rated 1 | 27 | 25
  Esthetic Anatomical Form at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Esthetic Anatomical Form at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Esthetic Anatomical Form at end of study : Number of teeth rated 2 | 1 | 2
  Esthetic Anatomical Form at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Esthetic Anatomical Form at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Esthetic Anatomical Form at end of study : Number of teeth rated 3 | 0 | 0
  Esthetic Anatomical Form at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Esthetic Anatomical Form at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Esthetic Anatomical Form at end of study : Number of teeth rated 4 | 0 | 0
  Esthetic Anatomical Form at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Esthetic Anatomical Form at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Esthetic Anatomical Form at end of study : Number of teeth rated 5 | 0 | 0

2. Primary Outcome: Change in Functional Properties: Number of Teeth, Rated 1 (Most Desirable Outcome) to 5 (Least Desirable Outcome), in Each Functional Category
Description: The following properties will be evaluated using the Hickel Grading Criteria:
  1. Fracture of material and retention
  2. Marginal adaptation
  3. Approximate anatomical form - contact point
  4. Radio-graphic examination (when applicable)
  5. Patient's view
  Each criteria will be graded by blinded examiner in 5 point scale from 1 being excellent to 5 being clinically unacceptable
Time Frame: From Baseline up to 2 Years After Restoration Placement
Population: as for outcome 1
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | SonicFill™ 2 | Filtek™ Supreme
Number analyzed (Participants) | 45 | 45
Number analyzed (Teeth) | 45 | 45
Teeth
  Fracture of Material and Retention at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Fracture of Material and Retention at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Fracture of Material and Retention at end of study : Number of teeth rated 1 | 27 | 26
  Fracture of Material and Retention at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Fracture of Material and Retention at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Fracture of Material and Retention at end of study : Number of teeth rated 2 | 0 | 1
  Fracture of Material and Retention at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Fracture of Material and Retention at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Fracture of Material and Retention at end of study : Number of teeth rated 3 | 1 | 0
  Fracture of Material and Retention at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Fracture of Material and Retention at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Fracture of Material and Retention at end of study : Number of teeth rated 4 | 0 | 0
  Fracture of Material and Retention at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Fracture of Material and Retention at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Fracture of Material and Retention at end of study : Number of teeth rated 5 | 0 | 0
  Marginal Adaptation at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Marginal Adaptation at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Marginal Adaptation at end of study : Number of teeth rated 1 | 23 | 25
  Marginal Adaptation at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Marginal Adaptation at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Marginal Adaptation at end of study : Number of teeth rated 2 | 5 | 2
  Marginal Adaptation at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Marginal Adaptation at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Marginal Adaptation at end of study : Number of teeth rated 3 | 0 | 0
  Marginal Adaptation at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Marginal Adaptation at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Marginal Adaptation at end of study : Number of teeth rated 4 | 0 | 0
  Marginal Adaptation at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Marginal Adaptation at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Marginal Adaptation at end of study : Number of teeth rated 5 | 0 | 0
  Radiographic Examination at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Radiographic Examination at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Radiographic Examination at end of study : Number of teeth rated 1 | 26 | 26
  Radiographic Examination at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Radiographic Examination at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Radiographic Examination at end of study : Number of teeth rated 2 | 0 | 1
  Radiographic Examination at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Radiographic Examination at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Radiographic Examination at end of study : Number of teeth rated 3 | 2 | 0
  Radiographic Examination at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Radiographic Examination at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Radiographic Examination at end of study : Number of teeth rated 4 | 0 | 0
  Radiographic Examination at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Radiographic Examination at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Radiographic Examination at end of study : Number of teeth rated 5 | 0 | 0
  Patient's View at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Patient's View at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Patient's View at end of study : Number of teeth rated 1 | 27 | 27
  Patient's View at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Patient's View at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Patient's View at end of study : Number of teeth rated 2 | 0 | 0
  Patient's View at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Patient's View at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Patient's View at end of study : Number of teeth rated 3 | 1 | 0
  Patient's View at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Patient's View at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Patient's View at end of study : Number of teeth rated 4 | 0 | 0
  Patient's View at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Patient's View at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Patient's View at end of study : Number of teeth rated 5 | 0 | 0

3. Primary Outcome: Change in Biological Properties: Number of Teeth, Rated 1 (Most Desirable Outcome) to 5 (Least Desirable Outcome), in Each Biological Category
Description: The following properties will be evaluated using the Hickel Grading Criteria:
  1. Postoperative (hyper-)sensitivity and tooth vitality
  2. Recurrence of caries, erosion, abfraction
  3. Tooth integrity (enamel cracks, tooth fractures)
  4. Adjacent mucosa
  Each criteria will be graded by blinded examiner in 5 point scale from 1 being excellent to 5 being clinically unacceptable
Time Frame: From Baseline up to 2 Years After Restoration Placement
Population: as for outcome 1
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | SonicFill™ 2 | Filtek™ Supreme
Number analyzed (Participants) | 45 | 45
Number analyzed (Teeth) | 45 | 45
Teeth
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 1 | 27 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 2 | 1 | 0
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 3 | 0 | 0
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 4 | 0 | 0
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Postoperative (Hyper)-Sensitivity and Tooth Vitality at end of study : Number of teeth rated 5 | 0 | 0
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 1 | 27 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 2 | 1 | 0
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 3 | 0 | 0
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 4 | 0 | 0
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Recurrence of Caries, Erosion, Abfraction at end of study : Number of teeth rated 5 | 0 | 0
  Tooth Integrity at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Tooth Integrity at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 1 | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Tooth Integrity at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 2 | 0 | 0
  Tooth Integrity at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Tooth Integrity at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 3 | 0 | 0
  Tooth Integrity at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Tooth Integrity at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 4 | 0 | 0
  Tooth Integrity at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Tooth Integrity at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Tooth Integrity at end of study : Number of teeth rated 5 | 0 | 0
  Adjacent Mucosa at end of study : Number of teeth rated 1: number analyzed (Participants) | 29 | 29
  Adjacent Mucosa at end of study : Number of teeth rated 1: number analyzed (Teeth) | 28 | 27
  Adjacent Mucosa at end of study : Number of teeth rated 1 | 27 | 26
  Adjacent Mucosa at end of study : Number of teeth rated 2: number analyzed (Participants) | 29 | 29
  Adjacent Mucosa at end of study : Number of teeth rated 2: number analyzed (Teeth) | 28 | 27
  Adjacent Mucosa at end of study : Number of teeth rated 2 | 1 | 1
  Adjacent Mucosa at end of study : Number of teeth rated 3: number analyzed (Participants) | 29 | 29
  Adjacent Mucosa at end of study : Number of teeth rated 3: number analyzed (Teeth) | 28 | 27
  Adjacent Mucosa at end of study : Number of teeth rated 3 | 0 | 0
  Adjacent Mucosa at end of study : Number of teeth rated 4: number analyzed (Participants) | 29 | 29
  Adjacent Mucosa at end of study : Number of teeth rated 4: number analyzed (Teeth) | 28 | 27
  Adjacent Mucosa at end of study : Number of teeth rated 4 | 0 | 0
  Adjacent Mucosa at end of study : Number of teeth rated 5: number analyzed (Participants) | 29 | 29
  Adjacent Mucosa at end of study : Number of teeth rated 5: number analyzed (Teeth) | 28 | 27
  Adjacent Mucosa at end of study : Number of teeth rated 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 24 months.
Description: Other (Not Including Serious) Adverse Events: Adverse events that are not Serious Adverse Events.
Arm/Group | SonicFill™ 2 | Filtek™ Supreme
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 14/45 | 15/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SonicFill™ 2 (N=45) | Filtek™ Supreme (N=45)
Fracture of restorations (Product Issues) | 2 | 3
Soft tissue irritation (Skin and subcutaneous tissue disorders) | 3 | 3
Post operative sensitivity/Pain (Injury, poisoning and procedural complications) | 6 | 5
Pulp exposure risk, healing of non- study site, Alterantion of study site due to non-study site tx (General disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT03032705/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT03032705/ICF_001.pdf